CLINICAL TRIAL: NCT05796856
Title: Effect of Different Wavelengths of Repeated Low-Level Light Therapy on Choroidal and Retinal Blood Flow Among Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second People's Hospital of Foshan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: (2022)-0140
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Choroid; Retina

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repeated low-level light therapy (wavelength: 810 nm) (Experimental): Participants will be treated with repeated low level light therapy (wavelength of 650 nm) twice per weekday with an interval of at least 4 hours, each treatment last 3 minutes.
  Single-vision spectacles with power for correcting distance refraction will also be used if necessary.
  Interventions: Device: repeated low level light device (Eyerising [Suzhou Xuanjia Optoelectronics Technology)
- Repeated low-level light therapy (wavelength: 650 nm) (Active Comparator): Participants will be treated with repeated low level light therapy (wavelength of 650 nm) twice per weekday with an interval of at least 4 hours, each treatment last 3 minutes.
  Single-vision spectacles with power for correcting distance refraction will also be used if necessary.
  Interventions: Device: repeated low level light device (Eyerising [Suzhou Xuanjia Optoelectronics Technology)

INTERVENTIONS:
Device: repeated low level light device (Eyerising [Suzhou Xuanjia Optoelectronics Technology) — crossover device (repeated low level light device with wavelength of 810/650 nm- alternate to first group) Cross over arms after one month of use and one month of washout period.

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of different intensity of repeated low-level red-light (RLRL) therapy on the choroidal and retinal blood flow among adults.

DETAILED DESCRIPTION:
Repeated low-level red-light (RLRL) therapy is an emerging innovative and non-invasive treatment for a variety of eye diseases. Notably, RLRL was found to be effective in thickening choroidal thickness in a 1-year randomized controlled trial, indicating its potential in modulating blood flow in the fundus. However, it remains unclear how long it takes for the RLRL to make a difference in fundus blood flow and whether there is a dose-response.

The purpose of this study is to evaluate the different wavelengths of of repeated low level light therapy on the choroidal and retinal blood flow among adults. This study will be conducted with a randomized cross-over design with a total follow-up of 3 months. The repeated low level light therapy will be carried out in the study site under supervision according to a standard protocol. Detailed ophthalmic examinations, including visual acuity, intraocular pressure, optical coherence tomography/angiography, optical coherence tomography angiography, cycloplegic spherical equivalent refraction, slit lamp, and biological parameters will be evaluated at enrollment and during follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-40 years at enrolment.
2. Healthy adults with best corrected visual acuity equal to or better than 1.0 in both eyes.
3. Provision of consent and able to participate in all required activities of the study.

Exclusion Criteria:

1. Secondary myopia, such as a history of retinopathy of prematurity or neonatal problems, or syndromic myopia with a known genetic disease or connective tissue disorders, such as Stickler or Marfan syndrome; or high myopia < -8 diopters.
2. Strabismus and vision abnormalities (astigmatism > 3.5 D) in either eye.
3. Refractive media opacity: corneal opacities, cataracts, or implanted intraocular lens, etc.
4. Ocular abnormalities that affect retinal function: macular degeneration, diabetic retinopathy, retinal detachment, glaucoma, or ocular hypertension, endophthalmitis, uveitis, optic neuropathy, etc.
5. Previous history of refractive surgery, intraocular surgery, laser therapy, and intravitreal injection, etc.
6. Systemic abnormalities: diabetes, hypertension, etc.
7. Drugs therapies with toxicity effects on the retina: hydroxychloroquine, etc.
8. Prior treatment of myopia control in the past three months including drugs, orthokeratology, progressive addition lenses, bifocal lenses, etc.
9. Other contraindications, including but not limited to ocular or other systemic abnormalities, that the physician may consider inappropriate for enrolment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-08 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
1. Changes of macular choroidal thickness | 1 month
  Changes in the macular choroidal thickness are characterized as the difference following 1 month with RLRL therapy relative to the baseline which is measured by optical coherence tomography

SECONDARY OUTCOMES:
Changes in OCTA-derived parameters of choriocapillaris | 1 month
  Changes in the choriocapillaris microvasculature are characterized as the difference following 1 month with RLRL therapy relative to the baseline which is measured by optical coherence tomography angiography
Changes in OCTA-derived parameters of retina | 1 month
  Changes in retinal microvasculature are characterized as the difference following 1 month with RLRL therapy relative to the baseline which is measured by optical coherence tomography angiography
Incidence of treatment-emergent adverse events | 1 month
  Incidence of treatment-emergent adverse events is the rate of treatment-emergent adverse events over a specified period for subjects in the intervention arm. Subjects are asked to report any treatment-emergent adverse events, including but not limited to glare, flash blindness, and afterimages

IPD SHARING:
Plan to Share IPD: No